CLINICAL TRIAL: NCT04961203
Title: Pathways of Patients Followed in Palliative Care at the University Hospital of Strasbourg During the Year 2020: a Retrospective Pilot Study
Brief Title: Pathways of Patients Followed in Palliative Care at the University Hospital of Strasbourg: a Retrospective Pilot Study
Acronym: Palliatif
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8295
Record Dates: First submitted 2021-06-01; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: Palliative care; Pathways
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In view to develop a study design for a study that would analyze the pathways of palliative care prospectively, this work will identify the individual factors that would be significantly associated with typical pathways of palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Patient met by the palliative care mobile team or admitted in palliative care unit
* Patient who died between January 2020 and December 2020.

Exclusion Criteria:

* Minors and incapacitated adults, or deprived of liberty
* Patient who explained their disagreement with the use of medical data for research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient met by the palliative care mobile team or admitted in palliative care unit and who died between January 2020 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective study describing the patient care pathway | The files analyzed retrospectively concern the period from January 01, 2020 to December 31, 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Calvel, MD, PhD, Study Director — Service de soins Palliatifs - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de soins Palliatifs - Hôpitaux Universitaires de Strasbourg, Strasbourg, France